CLINICAL TRIAL: NCT03264417
Title: Pulmonary Function Test Study - Automated Interpretation
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: University Hospital, Ghent (Other); AZ Sint-Jan AV (Other); Ziekenhuis Oost-Limburg (Other); Jessa Hospital (Other); Onze Lieve Vrouwziekenhuis Aalst (Other); Centre Hospitalier Universitaire de Charleroi (Other); University Hospital St Luc, Brussels (Other); Centre Hospitalier Universitaire Saint Pierre (Other); University of Liege (Other); Centre Hospitalier du Luxembourg (Other); Maastricht University Medical Center (Other); University Medical Center Nijmegen (Other); University Medical Center Groningen (Other); University Hospital, Paris (Other); University Hospital, Grenoble (Other); Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Wim Janssens, Prof. Dr., KU Leuven
Other Study IDs: S60619
Record Dates: First submitted 2017-08-01; First posted 2017-08-29 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A multicentric study to explore variability when clinicians are intrepreting lung function tests. Comparison with results of in-house built software for automatic interpretation.

DETAILED DESCRIPTION:
This is a multi-center non-interventional retrospective study that will use data obtained from clinical routine. In the hospital, subjects with or without respiratory complaints undergo subset of (or complete) pulmonary function tests if clinically indicated. Results of these tests, expressed as numerical values are send to the clinical workstation (KWS) for immediate clinical use. These results are subsequently being interpreted by a clinician.

A random sample of 50 lung function printouts of subjects followed at the Leuven pulmonary service with a final diagnosis of a respiratory disease have been randomised. These anonymized printouts will be given to different pulmonologists for examination in 18 different centers and compared with the interpretation of in-house developed software.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years
2. Completed one or more pulmonary function tests

Exclusion Criteria:

1. Younger than 18
2. Lung transplantation, lung cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with or without respiratory complaints undergo subset of (or complete) pulmonary function tests
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Interclass correlation coëfficiënt for whole group | 6 months
  Variation in preferred primary diagnosis of respiratory disease given by every physician for every case (selection of one diagnosis out of a fixed panel of 9 possible diagnoses).

SECONDARY OUTCOMES:
Interclass correlation coëfficiënt for every case | 6 months
  Variation in preferred primary diagnosis of respiratory disease given by every physician for an individual case (selection of one diagnosis out of a fixed panel of 9 possible diagnoses).
Accuracy of physicians expressed as a percentage of correct diagnoses per case (%) | 6 months
  Comparison of diagnostic labels per case provided by the physicians with gold standard diagnosis based on clinical characteristics, complete pulmonary function test data and all other investigations (CT scan, biochmestry, functional test, biopsy, etc...) needed to come to a gold standard diagnosis.
Accuracy of physicans expressed as a percentage of correct diagnoses in total group (%) | 6 months
  Comparison of diagnostic labels per case provided by the physicians with gold standard diagnosis based on clinical characteristics, complete pulmonary function test data and all other investigations (CT scan, biochmestry, functional test, biopsy, etc...) needed to come to a gold standard diagnosis.
Accuracy of physicians expressed as a percentage of correct diagnoses per hospital (group) (%) | 6 months
  Comparison of diagnostic labels per case provided by the group of physicians per hospital with gold standard diagnosis based on clinical characteristics, complete pulmonary function test data and all other investigations (CT scan, biochmestry, functional test, biopsy, etc...) needed to come to a gold standard diagnosis.
Accuracy of software expressed as a percentage of correct diagnoses in total group, per hospital and per case | 6 months
  Comparing labels of in-house developed software for the clinical interpretation and diagnostic labeling of complete pulmonary function tests with GOLD standard based on all additional tests
Comparison of accuracy (% of correct diagnoses) of physicians with software | 6 months
  Comparing the diagnostic labels provided by in-house developed software for the clinical interpretation and diagnostic labeling of complete pulmonary function tests with those of physicans (in total group, per hospital and per case)

CONTACTS AND LOCATIONS:
Overall Officials: Wim Janssens, Prof. Dr., Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium